CLINICAL TRIAL: NCT04186442
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase I Clinical Trial to Compare the Safety and Efficacy of Botulax® Versus Botox® in Patient With Overactive Bladder
Brief Title: Evaluate the Safety and Efficacy of Botulax® Versus Botox® in Patient With Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-BOTOAB-PI-01
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin type A (Botulax®) (Experimental)
  Interventions: Drug: Botulinum toxin type A injection
- Botulinum toxin type A (Botox®) (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]

INTERVENTIONS:
Drug: Botulinum toxin type A injection — Experimental
  Other Names: Botulax®
  Arms: Botulinum toxin type A (Botulax®)
Drug: Botulinum Toxin Type A Injection [Botox] — Active Comparator
  Other Names: Botox®
  Arms: Botulinum toxin type A (Botox®)

SUMMARY:
To determine the efficacy and safety of Botulax® in treatment of Overactive Bladder

DETAILED DESCRIPTION:
A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase I Clinical Trial to Compare the Safety and Efficacy of Botulax® versus Botox® in Patient with Overactive Bladder

ELIGIBILITY:
Inclusion Criteria:

1. Female at the age of 19 or older
2. Subjects who agree to participate in the clinical study and voluntarily sign the written informed consent form
3. Subjects with idiopathic overactive bladder who meets the following conditions:

   1. Subjects with persistent overactive bladder symptoms for the last 12 weeks
   2. Subjects who are not properly controlled by the administration of anticholinergic agents for 4 weeks or more or who are difficult to treat due to adverse reactions
   3. Subjects with urinary incontinence, urgency, and urinary frequency symptoms
4. Subjects who are willing to perform clean intermittent catheterization (CIC), if needed

Exclusion Criteria:

Subjects who are eligible for any of the following conditions may not participate in this study:

1. Subjects with the following comorbidities:

   1. Subjects with peripheral motor neuron disease (eg. amyotrophic lateral sclerosis, motor neuropathy) or systemic neuromuscular junction disorders (eg. myasthenia gravis, Lambert-Eaton syndrome)
   2. Overactive bladder patients due to neurological factors (eg stroke, spinal cord disease, Parkinson's disease, etc.)
   3. Subjects with clinically significant stress incontinence
   4. Subjects with Urinary Tract Infections*

      * Culture showing ≥10^5 colony-forming units (CFU)/mL and leukocytes ≥5 high power field (HPF)
   5. Patients with acute urinary retention, or with a history or accompanying diseases that can cause urinary retention (urolithiasis, acute cystitis, foreign body in the bladder, bladder flow, etc.)
   6. Uncontrolled diabetes patients who meet one or more of the following criteria:

      * HbA1c ≥ 9% at screening
      * Patients with over 10 years of diabetes
      * Have diabetic chronic complications (eg diabetic neuropathy, diabetic nephropathy, diabetic retinopathy, etc.)
      * Patients taking a drug that causes glycosuria (sodium-glucose co-transporter 2 inhibitor, SGLT2 inhibitor)
2. Those who have had lower urinary tract surgery within 24 weeks before screening
3. Those who received botulinum toxin due to urinary system disease within 24 weeks before screening
4. Those who have been administered botulinum toxin type A within 12 weeks prior to screening or botulinum toxin type B within 16 weeks of treatment, or planned during the clinical trials
5. Those who have received or plan to receive oral medications for overactive bladder including anticholinergic drugs within 1 week prior to randomization
6. Those who received antiplatelet and anticoagulants within 1 week prior to randomization
7. Subjects with a history of hypersensitivity reactions to any of the components of the investigational product
8. Women of childbearing potential who are planning to become pregnant during the clinical trials or are not using an appropriate method of contraception
9. Those who participated in another clinical trial within 12 weeks prior to screening and received investigational product/medical device/medical procedure
10. Those who are sensitive to cephalosporin or penicillin antibiotics

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence rates | 12 weeks (during the clinical trial)
  To assess severity and frequency of reported TEAE (treatment-emergent adverse event), ADR (adverse drug reaction), and SAE (serious adverse event) after investigational product injection

SECONDARY OUTCOMES:
Urinary incontinence rate | Baseline to Week 2, Week 6, Week 12
  The change in the average number of Urinary incontinence per day at 2, 6 and 12 weeks from baseline
Voiding frequency rate | Baseline to Week 2, Week 6, Week 12
  The change in the average number of voiding frequency per day at 2, 6 and 12 weeks from baseline
Urinary urgency rate | Baseline to Week 2, Week 6, Week 12
  The change in the average number of urinary urgency (Urgency Rating Scale; URS≥2)per day at 2, 6 and 12 weeks from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, Korea, South Korea